CLINICAL TRIAL: NCT02972333
Title: Open Label, Multi-center, Prospective Study to Investigate the Efficacy and Safety of AZD9291 in Brain Metastases From Patients With EGFR T790M Positive NSCLC Who Have Received Prior Therapy With an EGFR-TKI
Brief Title: Open Label, Prospective Study to Investigate Efficacy and Safety of AZD9291 in BM From NSCLC Patients With EGFR T790M
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jinming Yu, Dean, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APOLLO
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: EGFR-TKI Resistant Mutation; Nonsmall Cell Lung Cancer; AZD9291; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — osimertinib; Radiotherapy; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD9291 80mg oral each day±RT (Experimental): AZD9291(80mg, QD, p.o.) was provided to patients with confirmed EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI and concurrent with brain metastasis. Radiation therapy will be implemented according to investigator's clinical practice(A 7-10 days washout period before radiotherapy and 1 week period after completion of brain radiothearpy before re-starting AZD9291.).
  Interventions: Drug: AZD9291 80mg oral each day; Radiation: Radiation therapy

INTERVENTIONS:
Drug: AZD9291 80mg oral each day — All eligible patients will have access to AZD9291 regimen through the ASTRIS study as long as they continue to show clinical benefit.
  Other Names: AZD9291, 80mg, QD, p.o. (2nd line or later)
Radiation: Radiation therapy — Radiation therapy will be implemented according to investigator's clinical practice.Based on the guidelines provided for the interruption of ADZ9291 with brain radiation therapy, a 7-10 days washout period before radiotherapy and 1 week period after completion of brain radiothearpy before re-starting AZD9291.
  Other Names: WBRT or SRS

SUMMARY:
The study aims to investigate the efficacy and safety of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI.

DETAILED DESCRIPTION:
Patients with confirmed EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI and concurrent with brain metastasis will be enrolled into the study. All eligible patients will have access to AZD9291 regimen through the ASTRIS study as long as they continue to show clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
2. Metastatic (stage IV) EGFRm NSCLC, not amenable to curative surgery or radiotherapy, with confirmation of the presence of the T790M mutation.
3. For patients with LM: Confirmed diagnosis of LM by positive CSF cytology. Diagnosis by MRI only is not eligible for study entry. At least one site of CNS leptomeningeal disease that can be assessed by magnetic resonance imaging (MRI) and which is suitable for repeat assessments. Measurable CNS or extracranial disease is not required.
4. For patients with measurable BM but without LM: At least one measurable intracranial lesion that, if previously irradiated, has progressed or not responded to radiation therapy, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter by magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements. Measurable extracranial disease is not required.
5. Prior therapy with an EGFR-TKI. Patients may have also received additional lines of treatment.
6. World Health Organization (WHO) performance status 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 3 months.
7. Adequate bone marrow reserve and organ function as demonstrated by complete blood count, biochemistry in blood and urine at baseline.
8. ECG recording at baseline showing absence of any cardiac abnormality as per exclusion criterion #10.
9. Female patients of childbearing potential must be using adequate contraceptive measures (see Restrictions, Section 3.5), must not be breast feeding, and must have a negative pregnancy test prior to start of dosing. Otherwise, they must have evidence of nonchild bearing potential as defined below:

   1. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   2. Women less than 50 years would be consider post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
   3. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
10. Male patients must be willing to use barrier contraception, i.e., condoms.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Previous (within 6 months) or current treatment with AZD9291
2. Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of AZD9291) any treatment known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A4 (Appendix B)
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, active infection* including hepatitis B, hepatitis C and human immunodeficiency virus, or significantly impaired bone marrow reserve or organ function, including hepatic and renal impairment, which in the investigator's opinion would significantly alter the risk/benefit balance.

   * active infection will include any patients receiving intravenous treatment for any infection and patients with hepatitis B or C surface antigen (+) - Patients receiving oral antiviral suppressive therapy for hepatitis B or C will be permitted to enrol in the study.
4. Patient with symptomatic central nervous system (CNS) metastases who is neurologically unstable or has required increasing doses of steroids to manage CNS symptoms within the 2 weeks prior to start AZD9291 administration.
5. Prior whole brain radiation therapy.
6. Known intracranial hemorrhage which is unrelated to tumor.
7. For patients with LM and/or BM, CNS complications that require urgent neurosurgical intervention (e.g. resection or shunt placement).
8. For patients with LM, inability to undergo collection of CSF.
9. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
10. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTcF) > 470 ms using Fredericia's formula :
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
11. Any unresolved toxicity from prior therapy CTCAE > grade 3 at the time of starting treatment
12. History of hypersensitivity to excipients of AZD9291 or to drugs with a similar chemical structure or class to AZD9291
13. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count < 1.5 x 10^9/L
    * Platelet count < 100 x 10^9/L
    * Haemoglobin < 90 g/L
    * Alanine aminotransferase > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
    * Aspartate aminotransferase > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
    * Total bilirubin > 1.5 times ULN. Total bilirubin >3 times the ULN in patients with documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or in the presence of liver metastases
    * Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by Cockcroft and Gault equation). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
    * If bone metastases are present and liver function is otherwise considered adequate by the investigator then elevated ALP will not exclude the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
PFSo (overall progression free survival) | 2 years
  To assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI by PFSo

SECONDARY OUTCOMES:
PFSe (extracranial progression-free survival) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
PFSi (intracranial progression-free survival) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
ORRo (overall objective response rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
ORRe (extracranial objective response rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
ORRi (intracranial objective response rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DCRo (overall disease control rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DCRe (extracranial disease control rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DCRi (intracranial disease control rate) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DoRo (overall duration of response) | 3 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DoRe (extracranial duration of response) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
DoRi (intracranial duration of response) | 2 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
OS(overall survival) | 3 years
  To further assess the efficacy of AZD9291 in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI in pre-specified patient subgroups, e.g. AZD9291 single regimen, AZD9291 (before or after radiotherapy) with radiotherapy etc.
Adverse events/Serious adverse events | 2 years
  To evaluate the safety and tolerability profile of AZD9291 and subgroups such as AZD9291 single regimen, AZD9291(before or after radiotherapy) with radiotherapy and etc. in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI.
QoL | 2 years
  To assess disease-related symptoms and QoL in overall population as well as in pre-specified subgroups, e.g. AZD9291 single regimen, AZD9291(before or after radiotherapy) with radiotherapy etc. in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI.
Cognitive function | 2 years
  To assess disease-related symptoms and cognitive function in overall population as well as in pre-specified subgroups, e.g. AZD9291 single regimen, AZD9291(before or after radiotherapy) with radiotherapy etc. in brain metastases from patients with EGFR T790M positive NSCLC who have received prior therapy with an EGFR-TKI.

OTHER OUTCOMES:
T790M mutation positive rate | 2 years
  To investigate the effect of AZD9291 on the inhibition of proof of mechanism biomarkers (to include, but not limited to EGFR T790M) in cell pellets from pre- and post-treatment CSF samples in comparison with blood samples.
Concordance of T790M status between CSF and plasma | 2 years
  To investigate the effect of AZD9291 on the inhibition of proof of mechanism biomarkers (to include, but not limited to EGFR T790M) in cell pellets from pre- and post-treatment CSF samples in comparison with blood samples.
Change of imputed ctDNA concentration before and after treatment | 2 years
  To investigate the effect of AZD9291 on the inhibition of proof of mechanism biomarkers (to include, but not limited to EGFR T790M) in cell pellets from pre- and post-treatment CSF samples in comparison with blood samples.
Proportion of each genetic mutation | 2 years
  To investigate the effect of AZD9291 on the inhibition of proof of mechanism biomarkers (to include, but not limited to EGFR T790M) in cell pellets from pre- and post-treatment CSF samples in comparison with blood samples.
Change from baseline in glucose and protein levels | 2 years
  To evaluate the changes from baseline in CSF biochemistry to support the demonstration of the anti-tumour effect of AZD9291 in addition to CSF cytology.
Change from baseline in tumor cell count | 2 years
  To evaluate the changes from baseline in CSF biochemistry to support the demonstration of the anti-tumour effect of AZD9291 in addition to CSF cytology.
AZD9291 concentration level in CSF/plasma | 2 years
  To explore potential relation between relevant efficacy measures, biomarkers or safety variables and plasma or CSF concentration of AZD9291 (or metabolites).

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, MD.PhD., Principal Investigator — Shandong Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xing L, Pan Y, Shi Y, Shu Y, Feng J, Li W, Cao L, Wang L, Gu W, Song Y, Xing P, Liu Y, Gao W, Cui J, Hu N, Li R, Bao H, Shao Y, Yu J. Biomarkers of Osimertinib Response in Patients with Refractory, EGFR-T790M-positive Non-Small Cell Lung Cancer and Central Nervous System Metastases: The APOLLO Study. Clin Cancer Res. 2020 Dec 1;26(23):6168-6175. doi: 10.1158/1078-0432.CCR-20-2081. Epub 2020 Aug 17. PMID 32817079